CLINICAL TRIAL: NCT01096069
Title: Expressão de Cregs e a Resposta clínica em Pacientes AR Tratada Com Rituximabe
Brief Title: Complement Regulatory Proteins Expression and Clinical Response in Rheumatoid Arthritis (RA) Patients Treated With Rituximab
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Ricardo Machado Xavier, Hospital de Clinicas de Porto Alegre
Other Study IDs: 09/585
Record Dates: First submitted 2010-02-23; First posted 2010-03-30 (Estimated); Last update posted 2010-03-30 (Estimated); Status verified 2010-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rituximab, rheumatoid arthritis, CD55, CD59
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Rituximab: Rheumatoid arthritis patients undergoing treatment with rituximab.

SUMMARY:
There is a correlation between the CD55, CD59, CD35 and CD46 expression on B lymphocytes of patients before and after treatment with rituximab and the level of depletion and repopulation time for these cells. The theoretical rationale of the study assumes that the correlation, if any, will be a negative correlation. However, the hypothesis of positive correlation (two-tailed test) will also be tested.

DETAILED DESCRIPTION:
Rituximab, an anti-CD20 monoclonal antibody, is a new alternative treatment for patients with severe immune diseases and resistance to conventional treatment. One of the mechanisms of action of this drug is the complement-mediated lysis. Most RA patients respond well to rituximab treatment, however, some are refractory and mechanism of this non-response is still unclear. The role of CD55 and CD59 protein and its overexpression as a mechanism of resistance to rituximab treatment in lymphoma patients have been investigated. However, there has not been studied a correlation between the intensity of expression of these regulatory molecules on B cells of RA patients and resistance to treatment with Rituximab.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both gender, aged greater than or equal to 18 years; and lower than 70 years.
2. Patients diagnosed with RA for at least 6 months according to the criteria of the American College of Rheumatology (ACR) in 1987 for classification of AR.
3. Patients with a medical indication for therapy with rituximab, with prescription of this therapy for the first time and have not yet received the first dose.
4. DAS28 score greater than or equal to 3.2.
5. Use of adequate contraception, as judged from the attending physician.
6. Desire to participate voluntarily, the ability to understand the protocol, documented by signing the consent form (attached).

Exclusion Criteria:

1. overlapping rheumatic disease, autoimmune lymphoproliferative and neoplastic.
2. active infection, patients with the use of cytotoxic drugs, presence of positive serology for HCV, HBV and HIV, active or latent tuberculosis.
3. allergy or hypersensitivity to rituximab.
4. pregnant woman or performing breastfeeding.
5. participating in another clinical study with intervention.
6. with functional class IV defined based on the criteria of Steinbrocker functional classification for RA.
7. prior therapy with Rituximab.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with RA and clinical indication for treatment with rituximab and who have obtained access to medication (private purchase, delivery by a private health plan, lawsuit or donation by the laboratory Roche) will be invited to participate in the study during the physician appointment.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2010-06; Primary Completion 2010-12 (Estimated); Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo M Xavier, PhD, Study Director — HCPA